

Title: An Open-Label, Single-center, Parallel, Phase 1 Study to Determine the Pharmacokinetics of Single- and Multiple- Oral Doses of TAK-438 10 mg and 20 mg in Healthy Adult Chinese

NCT Number: NCT03085836

SAP Approve Date: 30 August 2017

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.



#### STATISTICAL ANALYSIS PLAN

STUDY NUMBER: TAK-438\_114

An Open-Label, Single-center, Parallel, Phase 1 Study to Determine the Pharmacokinetics of Single- and Multiple- Oral Doses of TAK-438 10 mg and 20 mg in Healthy Adult Chinese Subjects

#### PHASE 1

Version: Final 2
Date: 30 August 2017

| Prepared | by: |
|----------|-----|
|----------|-----|

PPD

#### Based on:

Protocol Version: Amendment 02 Protocol Date: 21 December 2016

#### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda

## 1.1 Approval Signatures

Electronic signatures can be found on the last page of this document.

**Study Title:** An Open-Label, Single-center, Parallel, Phase 1 Study to Determine the

Pharmacokinetics of Single- and Multiple- Oral Doses of TAK-438 10 mg

and 20 mg in Healthy Adult Chinese

| A | n | n | r | n | v | ล | ls | • |
|---|---|---|---|---|---|---|----|---|
| | ν | μ | | v | • | a | 13 | ۰ |

| PPD | Date |
|-----|------|
| PPD | Date |
| PPD | Date |
| PPD | Date |
| PPD | Date |

| 2.0 | TABLE OF CO | ONTENTS | |
|---|---|---|---|
| 1 | .1 Approval Sig | gnatures | 2 |
| 2.0 | TABLE OF CO | NTENTS | 3 |
| L | ist of In-Text Table | es | 4 |
| L | ist of In-Text Figur | res | 4 |
| 3.0 | LIST OF ABBR | EVIATIONS | 5 |
| 4.0 | OBJECTIVES | | 7 |
| 4 | .1 Primary Obj | ectives | 7 |
| 4 | .2 Secondary O | Objectives | 7 |
| 4 | .3 Additional C | Objectives | 7 |
| 4 | .4 Study Design | n | 7 |
| 5.0 | ANALYSIS EN | DPOINTS | 9 |
| 5 | .1 Primary End | points | 9 |
| 5 | .2 Additional E | indpoints | 10 |
| 6.0 | DETERMINAT | ION OF SAMPLE SIZE | 11 |
| 7.0 | METHODS OF | ANALYSIS AND PRESENTATION | 12 |
| 7 | .1 General Prin | ciples | 12 |
| | 7.1.1 Study De | efinitions | 12 |
| | 7.1.2 Definitio | n of Study Days | 12 |
| | 7.1.3 Definitio | n of Study Visit Windows | 12 |
| | | of Data Conversion and Handling of Missing Data | |
| 7 | .2 Analysis Set | S | 14 |
| 7 | .3 Disposition of | of Subjects | 14 |
| | • | formation | |
| | 7.3.2 Screen F | ailures | 14 |
| | • | Eligibility | |
| | • | on of Subjects | |
| | | Deviations and Analysis Sets | |
| 7 | • 1 | c and Other Baseline Characteristics | |
| 7 | | tory and Concurrent Medical Conditions | |
| | | History and Concomitant Medications | |
| | • | alysis | |
| 7 | | netic/Pharmacodynamic Analysis | |
| | | okinetic Analysis | |
| | 7 8 2 Pharmac | odynamic Analysis | 19 |

Schematic of Study Design ......8

Figure 4.a

#### 3.0 LIST OF ABBREVIATIONS

AE adverse event

Ae<sub>t</sub> amount of drug excreted in urine from time 0 to time t
Ae<sub>t</sub> amount of drug excreted in urine during a dosing interval

aPTT activated partial thromboplastin time

 $AUC_{\infty}$  area under the plasma concentration-time curve from time 0 to infinity  $AUC_{\tau}$  area under the plasma concentration-time curve during a dosing interval

 $AUC_{\tau,ss}$  area under the plasma concentration-time curve during a dosing interval, at steady

state

BID twice daily
BMI body mass index

CFDA China Food and Drug Administration

CL<sub>R</sub> renal clearance

C<sub>max</sub> maximum observed plasma concentration

C<sub>max.ss</sub> maximum observed plasma concentration, at steady state

CRF case report form
CV coefficient of variation
CYP cytochrome P450
ECG electrocardiogram

f<sub>e t</sub> Fraction of administered dose of drug excreted in urine from time 0 to time t.

Molecular weight adjustment needed for metabolites

 $f_{e,\tau}$  Fraction of administered dose of drug excreted in urine during a dosing interval.

Molecular weight adjustment needed for metabolites.

GGT γ-glutamyl transferase

HDL high density lipoprotein

LDH lactate dehydrogenase

LDL low density lipoprotein

LLN lower limit of normal

MAV markedly abnormal values

Medical Dictionary for Regulatory Activities

PD pharmacodynamics
PK pharmacokinetics
PT Preferred Term
PT prothrombin time

PT/INR prothrombin time/international normalized ratio

PTE pretreatment event

QD once daily

QTcF QT interval corrected by Fridericia's method

SAP statistical analysis plan SOC System Organ Class TAK-438F freebase of TAK-438 TEAE treatment-emergent adverse event  $t_{1/2z}$  terminal disposition phase half-life  $t_{max}$  time of first occurrence of  $C_{max}$ 

 $t_{max,ss}$  time of first occurrence of  $C_{max}$ , at steady state

ULN upper limit of normal

WHO Drug World Health Organization Drug Dictionary

#### 4.0 OBJECTIVES

#### 4.1 Primary Objectives

The primary objective is to determine the pharmacokinetics of TAK-438 in healthy adult Chinese subjects after both single and multiple dose administration.

### 4.2 Secondary Objectives

Not applicable.

#### 4.3 Additional Objectives

#### 4.4 Study Design

This is a phase 1, parallel, open-label, single- and multiple-dose study of oral TAK-438 involving 36 healthy Chinese subjects between the ages of 18 and 45, inclusive, and considered eligible based on the inclusion and exclusion entry criteria.

Screening for potential subjects will occur between 28 and 2 days prior to confinement at the phase 1 unit. Selected eligibility criteria will be reconfirmed on Day -1 (Check In) prior to assignment to the 10 mg or 20 mg once daily or 20 mg twice daily cohort, predose blood and urine sampling for pharmacokinetic (PK) measurements will also be taken. Having fasted for a minimum of 10-hours a single oral dose of TAK-438 will be administered on Day 1 followed by a pharmacokinetic sampling period of 48 hours. On Days 3 through 9, subjects will receive their assigned daily dose(s) of TAK-438 followed by another pharmacokinetic sampling period of 48 hours (for subjects on a once daily regimen), or 12 hours (for those assigned to the 20 mg twice daily regimen). The subject will be confined to the phase 1 unit from Day -1 (Check-In) through to Day 11 (Check-Out) and will be contacted by the study site for a follow-up phone call on Day 18.

Besides monitoring concomitant medications and adverse events (AE), physical examination, electrocardiogram (ECG), vital signs and clinical laboratory tests will be conducted to monitor safety. A schematic of the study design is presented in Figure 4.a.

Figure 4.a Schematic of Study Design

| Screening | Period Treatment Period | | | | | Follow-Up | | |
|---|---|---|---|---|---|---|---|---|
| Screening | Check-<br>In | Single Dose/<br>PK | 48-hour<br>PK | Multiple<br>Dosing (a) | Dosing<br>and PK | 48-hour PK /<br>Observation | Check-<br>Out | Follow-up<br>Telephone<br>Visit |
| Days -28<br>to -2 | Day -1 | Day 1 | Day 2 | Days 3-8 | Day 9 | Day 10 | Day 11 | Day 18 ± 3<br>days |
| | | TAK-438<br>single dose 10<br>mg or 20 mg | de dose 10 10 mg or 20 mg or | | | | | |
| ← Confinement → | | | | | | | | |

PK=pharmacokinetic.

A summary of the dose cohorts is presented in Table 4.a.

 Table 4.a
 Summary of Dose Cohorts

| Cohort | TAK-438 Dose (shown as free base amount) | Subjects |
|--------|------------------------------------------|----------|
| 1 | TAK-438 10 mg once daily | 12 |
| 2 | TAK-438 20 mg once daily | 12 |
| 3 | TAK-438 20 mg twice daily | 12 |

A schematic of the dosing schedule and sampling, by cohort, is provided in Table 4.b.

 Table 4.b
 Schematic of Dosing and PK Sampling, by Cohort

| Regimen | Event | D1 | D2 | D3 | D4 | D5 | D6 | D7 | D8 | D9 | D10 | D11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 | Dosing | <b>1</b> | | $\uparrow$ | $\uparrow$ | $\uparrow$ | $\uparrow$ | $\uparrow$ | $\uparrow$ | $\uparrow$ | | |
| (10 mg QD) | PK sampling | <del></del> | | > | • | • | • | • | • | <del></del> | | > |
| Cohort 2 | Dosing | <b>↑</b> | | $\uparrow$ | $\uparrow$ | $\uparrow$ | $\uparrow$ | $\uparrow$ | $\uparrow$ | <b>↑</b> | | |
| (20 mg QD) | PK sampling | <del></del> | | > | • | • | • | • | • | <del></del> | | > |
| Cohort 3 | Dosing | $\uparrow$ | | $\uparrow \downarrow$ | $\uparrow \downarrow$ | $\uparrow \downarrow$ | $\uparrow \downarrow$ | $\uparrow \downarrow$ | $\uparrow \downarrow$ | $\uparrow \downarrow$ | | |
| (20 mg BID) | PK sampling | $\leftarrow$ | | > | • | • | • | • | • | $\leftrightarrow$ | | |

↑: Morning dose,; ↓: Evening dose; ↔: Serial PK; • Trough PK

#### 5.0 ANALYSIS ENDPOINTS

#### **5.1** Primary Endpoints

The Primary endpoints for this study are the pharmacokinetic parameters derived from the plasma and urine concentrations of TAK-438F and its metabolites M-I, M-II, M-III and M-IV-Sul assessed after the first dose on Day 1 and after the final repeat dose on Day 9 as required.

The following pharmacokinetic parameters will be calculated from plasma concentrations of TAK-438F, M-I, M-II, M-III and M-IV-Sul:

#### Day 1

- Maximum observed plasma concentration (C<sub>max</sub>).
- Time to reach  $C_{max}$  ( $t_{max}$ ).
- Area under the plasma concentration-time curve from time 0 to infinity (AUC $_{\infty}$ ).
- Area under the plasma concentration-time curve during a dosing interval (AUC $_{\tau}$ ).
- Terminal disposition half-life  $(t_{1/2z})$ .

#### Day 9

- Maximum observed plasma concentration, at steady state (C<sub>max,ss</sub>).
- Time to reach  $C_{max}$  at steady state  $(t_{max.ss})$ .
- Area under the plasma concentration-time curve during a dosing interval, at steady state (AUC<sub>τ.ss</sub>).

The following pharmacokinetic parameters will be calculated from urine concentrations of TAK-438F, M-I, M-II, M-III and M-IV-Sul:

#### <u>Day 1</u>

- Amount of drug excreted in urine from time 0 to time t (Ae<sub>t</sub>).
- Fraction of administered dose of drug excreted in urine from time 0 to time t (f<sub>e,t</sub>).
- Renal clearance (CL<sub>R</sub>).

#### Day 9

- Amount of drug excreted in urine during a dosing interval ( $Ae_{\tau}$ ).
- Fraction of administered dose of drug excreted in urine during a dosing interval  $(f_{e,\tau})$ .
- Renal clearance (CL<sub>R</sub>).

5.2 Additional Endpoints



#### 6.0 DETERMINATION OF SAMPLE SIZE

The sample size of 12 subjects per cohort is sufficient to evaluate the PK profile after single- and multiple-dose administration of TAK-438 10 mg and 20 mg. The sample size chosen for this study is based on precedent set by other pharmacokinetic studies of similar nature and guidelines issued by the China Food and Drug Administration (CFDA); it was not based on statistical considerations of power and sample size of TAK-438. The sample size is considered though to be sufficient for investigating the objectives of the study.

#### 7.0 METHODS OF ANALYSIS AND PRESENTATION

#### 7.1 General Principles

#### 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- TEAE: An AE whose date of onset occurs on or after the start of study drug. A TEAE whose relationship to study drug is missing will be considered drug-related. A TEAE whose intensity is missing will be considered severe.
- PTE: An AE whose date of onset occurs before the start of study drug.
- Significant TEAE: Any AEs (not including serious TEAEs) that led to an intervention, including withdrawal of drug treatment or significant additional concomitant therapy.
- Descriptive statistics: number of subjects with non-missing values, mean, standard deviation, maximum, minimum, and quartiles
- Duration of exposure to study medication (days): date of last dose of study medication date of first dose of study medication + 1
- QTcF interval (msec): QT interval (msec) / (RR interval (msec)/1000)<sup>0.33</sup> (rounded to the nearest whole number)
- Baseline values: The last evaluable observation (ie, non-missing) before the first dose of study medication. If no evaluable observation is obtained before the first dose, the baseline value will be missing.

#### 7.1.2 Definition of Study Days

Study Day: The day before the first dose of the study medication will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. Other study days are defined relative to Study Day 1, eg, the day 2 days prior to Study Day 1 is Day -2 and the day after Study Day 1 is Day 2.

#### 7.1.3 Definition of Study Visit Windows

7.1.3.1 Plasma Concentrations of TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul

For each time, all evaluable observation (ie, non-missing) obtained in the corresponding time interval will be used. If more than one observation lies within the same time window, the observation with the closest sampling time to the scheduled time will be used. If there are two observations equidistant to the scheduled time, the later observation will be used.

TAK-438\_114 Statistical Analysis Plan Final 1

Visit: Days 1 and 9

| | | Scheduled Time | Time Interval (min) |
|---|---|---|---|
| Visit | Time | (min) | Sampling Time |
| Days 1 and 9 | Pre-morning dose | 0 | -30 – 0 |
| | 0.25 hours post–morning dose | 15 | 10 – 20 |
| | 0.5 hours post–morning dose | 30 | 25 – 35 |
| | 0.75 hours post–morning dose | 45 | 40 – 50 |
| | 1 hour post–morning dose | 60 | 55 – 65 |
| | 1.5 hours post–morning dose | 90 | 85 – 95 |
| | 2 hours post–morning dose | 120 | 115 – 125 |
| | 3 hours post–morning dose | 180 | 175 – 185 |
| | 4 hours post–morning dose | 240 | 235 – 245 |
| | 6 hours post–morning dose | 360 | 355 – 365 |
| | 8 hours post–morning dose | 480 | 470 – 490 |
| | 10 hours post–morning dose | 600 | 590 - 610 |
| | 12 hours post–morning dose | 720 | 710 – 730 |
| | 16 hours post–morning dose* | 960 | 950 – 970 |
| | 24 hours post–morning dose* | 1440 | 1430 – 1450 |
| | 36 hours post–morning dose* | 2160 | 2150 – 2170 |
| | 48 hours post–morning dose* | 2880 | 2870 - 2890 |

<sup>\*</sup> Blood samples collection at these time points on Day 9 is not scheduled for Cohort 3, ie, subjects assigned to the 20 mg BID regimen.

Visit: Days 4-8

| | | <b>Scheduled Time</b> | Time Interval (min) |
|------------|------------------|-----------------------|---------------------|
| Visit | Time | (min) | Sampling Time |
| Days 4 - 8 | Pre-morning dose | 0 | -30 – 0 |

#### 7.1.3.2 Other Endpoints

The baseline visit is defined as the period before the first dose of study medication, and post-baseline visits are defined in line with CRF-recorded visits. The last evaluable observation (ie, non-missing) in the baseline visit will be used as the baseline value, and all evaluable observation will be used for each post-baseline visit.

#### 7.1.4 Method of Data Conversion and Handling of Missing Data

No imputation of missing data or of excluded data will be applied. Values below the lower limit of quantification will be handled as 0.

### 7.2 Analysis Sets

The safety analysis set used for primary analysis will consist of subjects who received at least 1 dose of the study drug.

The PK analysis set will consist of subjects who received the study drug, who have sufficient plasma/urine concentration data to calculate at least 1 pharmacokinetic parameter, and completed the minimum protocol specified procedures with no significant protocol deviations, which are listed below:

- Subjects who did not meet inclusion criteria #3, #4 or #5.
- Subjects who met exclusion criteria #1, #4, #6, #7, #8, #10, #11, #12, #13, #14, or #18.
- Subjects who have violated the rules specified in section 7.3 (excluded medications and dietary products) of the protocol up to 48 hours after the last dose on Day 9.
- Subjects who did not receive the study drug at some scheduled time of administration.

#### 7.3 Disposition of Subjects

#### 7.3.1 Study Information

Analysis Set: All Subjects Who Signed the Informed Consent Form
Analysis Variables: Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical Methods: (1) Study Information

Study information shown in the analysis variables section will be provided.

#### 7.3.2 Screen Failures

Analysis Set: All Subjects Who Did Not Enter the Treatment Period Analysis Variables: Age (years) [Min<= - <30, 30<= - <40, 40<= - <=Max]

Gender [Male, Female]

Race [American Indian or Alaska Native, Asian, Black or African American,

Native Hawaiian or Other Pacific Islander, White]

Analytical Methods: (1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for continuous

variables will be provided.

#### 7.3.3 Subject Eligibility

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Variables: Eligibility Status [Yes, No]

Primary Reason for Subject Not Being Eligible [Pretreatment Event/Adverse Event,

Significant Protocol Deviation,

Lost to Follow-Up, Voluntary Withdrawal, Study Termination,

Did Not Meet Entrance Criteria,

Other

Analytical Methods: (1) Eligibility for Entrance into the Treatment Period

Frequency distributions will be provided. When calculating the percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will be used as

the denominator.

#### 7.3.4 Disposition of Subjects

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis Variables: Study Drug Administration Status [No]

Reason for Not Being Treated [Pretreatment Event/Adverse Event,

Significant Protocol Deviation,

Lost to Follow-Up,

Voluntary Withdrawal, Study Termination,

Pregnancy, Other]

Study Drug Completion Status [Completed Study Drug,

Prematurely Discontinued Study Drug]

Reason for Discontinuation of Study Drug [Pretreatment Event/Adverse Event,

Significant Protocol Deviation,

Lost to Follow-Up,

Voluntary Withdrawal, Study Termination,

Pregnancy, Other]

Analytical Methods: (1) Disposition of Subjects

Frequency distributions will be provided for each cohort and overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation of study drug, the total number of subjects who prematurely discontinued

the study drug will be used as the denominator.

(2) Flow Chart of Subject Distribution

Flow chart will be provided.

### 7.3.5 Protocol Deviations and Analysis Sets

#### **Protocol Deviations**

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis Variables: Protocol Deviation [Entry Criteria, Concomitant Medication,

Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria

Analytical Methods: (1) Protocol Deviations

Frequency distribution will be provided by cohort and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be

counted only once.

**Analysis Sets** 

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis Variables: Analysis Sets

PK Analysis Set [Included] Safety Analysis Set [Included]

Analytical Methods: (1) Analysis Sets

Frequency distributions will be provided by cohort and overall.

#### **Demographic and Other Baseline Characteristics** 7.4

Analysis Set: PK Analysis Set

Safety Analysis Set

Analysis Variables: Age (years)  $[Min \le - <30, 30 \le - <40, 40 \le - <=Max]$ 

> Gender [Male, Female]

[American Indian or Alaska Native, Asian, Race

Black or African American.

Native Hawaiian or Other Pacific Islander,

White]

Height (cm)  $[Min \le - < 150, 150 \le - < 160,$ 

 $160 \le -170, 170 \le -180$ 

Weight (kg) (Baseline)  $[Min \le -.. \le 50.0, 50.0 \le -.. \le 60.0]$ 

 $60.0 \le -80.0$ ,  $70.0 \le -80.0$ ,

 $80.0 \le - \le Max$ 

BMI (kg/m<sup>2</sup>) (Baseline)  $Min \le - <19.0, 19.0 \le - <=24.0,$ 

 $24.0 < - \le Max$ 

**Smoking Classification** [The Subject Has Never Smoked,

The Subject Is a Current Smoker, The Subject Is an Ex-smoker]

Consumption of Alcohol [Drink Every day,

> Drink a Couple of Days Per Week, Drink a Couple of Days Per Month,

Never Drink]

Consumption of Caffeine [Yes, No]

[\*1/\*1, \*1/\*2, \*1/\*3, \*2/\*2, \*2/\*3, \*3/\*3] CYP2C19 Genotype

Analytical Methods: (1) Summary of Demographics and Other Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for continuous

variables will be provided by cohort and overall.

#### 7.5 **Medical History and Concurrent Medical Conditions**

Medical history is defined as significant conditions or diseases that stopped at or prior to the time of informed consent. Concurrent medical conditions are defined as significant conditions ongoing or present at the time of informed consent.

Medical history and concurrent medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, version 19.0) coding system.

There will be no analysis of medical history and concurrent medical conditions.

#### 7.6 **Medication History and Concomitant Medications**

Medication history information includes any medication relevant to eligibility criteria stopped prior to signing of informed consent. Concomitant medications are recorded on the eCRF and include any medications, other than the study drug, taken at any time between informed consent and on or prior to the last dose of study drug.

Medication history and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO Drug) version 2016Q1 or higher.

There will be no analysis of medication history and concomitant medications.

#### 7.7 Efficacy Analysis

Not applicable.

#### 7.8 Pharmacokinetic/Pharmacodynamic Analysis

#### 7.8.1 Pharmacokinetic Analysis

#### Plasma Concentrations of TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul

Analysis Set: PK Analysis Set

Analysis Variable: Plasma Concentrations of TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul

Time Point: Visit: Days 1 and 9

Pre-morning dose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16\*, 24\*, 36\*, 48\* hours post-morning dose (relative to start time of morning dose at Day 1 or 9)

\* Blood samples collection at these time points on Day 9 is not scheduled for Cohort 3,

ie, subjects assigned to the 20 mg BID regimen.

Visit: Days 4-8

Pre-morning dose (0 hours)

Analytical Methods: The following summaries will be provided for each analyte by cohort.

#### (1) Summary of Plasma Concentrations by Time Point

Descriptive statistics for observed values will be provided for each time point. In addition, geometric mean, and %CV will be provided

#### (2) Concentration-time Profiles for Individual Subjects

Observed values will be plotted using individual case plot.

#### (3) Mean Concentration-time Profiles with Standard Deviations

Mean of plasma concentration will be plotted by time point using linear scales and common

log scales for Days 1-9, Day 1 and Day 9 respectively.

Plasma PK Parameters of TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul

Analysis Set: PK Analysis Set

Analysis Visit and

Plasma PK Parameters of TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul

Variable:

Visit: Day 1

 $\begin{array}{ccc} C_{max} & & t_{max} & AUC_{\infty} \\ AUC_{\tau} & & t_{1/2z} & & \lambda_{z} \end{array}$ 

CL/F  $V_z/F$ 

Visit: Day 9

 $\begin{array}{ccc} C_{max,ss} & & t_{max,ss} & AUC_{\tau,ss} \\ t_{1/2z} & & \lambda_z & CL/F_{ss} \\ V_z/F_{ss} & & R_{ac(AUC)} & R_{ac(Cmax)} \end{array}$ 

Analytical Methods: The following summaries will be provided for each analyte by cohort.

(1) Summary of Plasma PK Parameters

Descriptive statistics for PK parameters will be provided. In addition, geometric mean and

%CV will be computed for  $C_{max}$  and AUCs.

Urine PK Parameters of TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul

Analysis Set: PK Analysis Set

Analysis Visit and Urine PK Parameters of TAK-438F, Its Metabolites M-I, M-II, M-III and M-IV-Sul, and the

Variable: Total of TAK-438F and Its Metabolites

Visit: Day 1

 $Ae_t$   $f_{e,t}$   $CL_R$ 

Visit: Day 9

 $Ae_{\tau}$   $f_{e,\,\tau}$   $CL_R$ 

Analytical Methods: The following summaries will be provided for each analyte by cohort.

(1) Summary of Urine PK Parameters

Descriptive statistics for PK parameters will be provided. Here, only fe will be summarized

for the total of TAK-438F and its metabolites.

#### 7.8.2 Pharmacodynamic Analysis

Not applicable.

#### 7.9 Other Outcomes

Not applicable.

#### 7.10 Safety Analysis

#### 7.10.1 Adverse Events

#### 7.10.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Variables: TEAE

Categories: Relationship to Study Drug [Related, Not Related]

Intensity [Mild, Moderate, Severe]

Analytical Methods: The following summaries will be provided for each cohort.

#### (1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 2) Relationship of Treatment-Emergent Adverse Events to Study Drug (number of events, number and percentage of subjects)
- 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 4) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)
- 5) Relationship to Study Drug of Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)
- 6) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 7) Relationship of Serious Treatment-Emergent Adverse Events to Study Drug (number of events, number and percentage of subjects)
- 8) Serious Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)
- 9) Treatment-Emergent Adverse Events Resulting in Death (number of events, number and percentage of subjects)
- 10) Significant Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 11) Relationship of Significant Treatment-Emergent Adverse Events to Study Drug (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

#### Number of subjects

- Summaries for 2), 5), 7) and 11)
  - A subject with occurrences of TEAE in both categories (ie, Related and Not Related) will be counted once in the Related category.
- Summary for 3)
  - A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.
- Summaries other than 2), 3), 5), 7) and 11)

## A subject with multiple occurrences of TEAE will be counted only once.

#### Number of events

For each summary, the total number of events will be calculated.

#### 7.10.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Variables: TEAE

Categories: Intensity [Mild, Moderate, Severe]

Analytical Methods: The following summaries will be provided using frequency distribution for each cohort.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by SOC only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Drug-Related Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (9) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (10) Serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (11) Significant Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (12) Drug-Related Significant Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

#### Number of subjects

- Summary tables other than (5), and (6)
  - A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (5) and (6)
  - A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.

7.10.1.3 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Variables: PTE

Analytical Methods: The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will

be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Pretreatment Events by System Organ Class and Preferred Term

(2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in

that PT.

### 7.10.2 Clinical Laboratory Evaluations

#### Hematology and Serum Chemistry

Analysis Set: Safety Analysis Set

Analysis Variables: Hematology

Red blood cells ( $\times 10^{12}$ /L) White blood cells ( $\times 10^{9}$ /L) Hemoglobin (g/L)

Hematocrit (%) Platelets ( $\times 10^9/L$ )

White blood cell differential (Neutrophils (%), Eosinophils (%), Basophils (%),

Monocytes (%), Lymphocytes (%))

PT/INR PT (sec) aPTT (sec)

Reticulocyte percentage

(%)

Serum Chemistry

Alanine aminotransferase Alkaline phosphatase (U/L) Aspartate aminotransferase

(U/L) (U/L)

GGT (U/L) Total bilirubin (µmol/L) Direct bilirubin (µmol/L)

Lactose dehydrogenase Creatine kinase (U/L) Albumin (g/L)

(U/L)

Total protein (g/L) Serum creatinine (umol/L) Blood urea (mmol/L)

Uric Acid (mmol/L) HDL Cholesterol (mmol/L) LDL Cholesterol (mmol/L)

Triglycerides (mmol/L) Glucose (mmol/L) Potassium (mmol/L)
Sodium (mmol/L) Magnesium (mmol/L) Calcium (mmol/L)

Chloride (mmol/L) Amylase (U/L)

Visit: Baseline, Days 3, 9 and 11.

Analytical Methods: The following summaries will be provided for each cohort. Liver function testing

measurements at local laboratories are not used for the summaries.

#### (1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - baseline) will be provided for each visit.

#### (2) Summary of Shifts of Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided. For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

# (3) Number and Percentage of Subjects with Markedly Abnormal Values of Laboratory Test results

Overall frequency distributions of MAV during treatment phase will be provided. If a laboratory test result has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### <u>Urinalysis</u>

Analysis Set: Safety Analysis Set

Analysis Variables : pH  $[Min \le -<5.0, 5.0 \le -<=8.5, 8.5 < -<=Max]$ 

Specific gravity  $[Min \le - <1.005, 1.005 \le - <=1.030, 1.030 < - <=Max]$ 

Protein [Negative, Positive]
Glucose [Negative, Positive]
Nitrites [Negative, Positive]
Bilirubin [Negative, Positive]
Ketones [Negative, Positive]
Urobilinogen [Normal, Abnormal]

Microscopic Analysis

RBC (/HPF) [Negative, Positive]
WBC (/HPF) [Negative, Positive]
Hyaline casts (/LPF) [Not Found, Positive]
Granular casts (/LPF) [Not Found, Positive]

Epithelial cells ( $\times 10^6$ /L) [Min<= - <2.0, 2.0<= - <=10.0, 10.0< - <=Max]

Visit: Baseline, Days 3, 9 and 11.

Analytical Methods: The following summaries will be provided for each cohort.

#### (1) Summary of Shifts of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

#### 7.10.3 Vital Signs

Analysis Set: Safety Analysis Set Analysis Variables: Body Temperature (°C)

> Systolic Blood Pressure (mmHg) Diastolic Blood Pressure (mmHg)

Respiratory Rate (bpm)

Pulse (bpm)

Visit: Baseline, Days 2-11

Analytical Methods: For each variable, following summary will be provided by cohort.

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit –

baseline) will be provided for each visit.

(2) Number and Percentage of Subjects with Markedly Abnormal Values of Vital Signs

**Parameters** 

Overall frequency distributions of MAV during treatment phase will be provided. If a vital sign parameter has both lower and upper MAV criteria, analysis will be performed for each.

Further details are given in Appendix.

#### 7.10.4 12-Lead ECGs

Analysis Set: Safety Analysis Set Analysis Variables: Heart Rate (bpm)

RR Interval (msec)
PR Interval (msec)
QT Interval (msec)
QTcF Interval (msec)
QRS Interval (msec)

12-Lead ECG Interpretation ["Within Normal Limits",

"Abnormal, Not Clinically Significant",

"Abnormal, Clinically Significant"]

Visit: Baseline, Days 1-11

Analytical Methods: For each variable other than 12-lead ECG interpretations, summary (1) will be provided by cohort.

For 12-lead ECG interpretations, summary (3) will be provided by cohort.

#### (1) Summary of ECG Parameters and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit – baseline) will be provided for each visit.

# (2) Number and Percentage of Subjects with Markedly Abnormal Values of ECG Parameters

Overall frequency distributions of MAV during treatment phase will be provided. If an ECG parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### (3) Summary of Shifts of ECG Parameters

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

#### 7.10.5 Other Observations Related to Safety

Not applicable.

#### 7.11 Interim Analysis

Not applicable.

#### 7.12 Changes in the Statistical Analysis Plan

From the SAP version 1.0, the following parts were updated. In 7.3.4, the subject flow chart was mentioned clearly. In 7.8.1, common log scales were applied to semi-log graphs for mean concentration-time profiles instead of natural log scales, and Ae was removed from the summary table for the total of TAK-438F and its metabolites. In 7.10.1.1 and 7.10.1.2, several tables for drug-related TEAEs were added. In 7.10.2, PT and microscopic analysis parameters were added to the analysis variables. In 9.1.1, the MAV criteria of blood urea was removed.

## 8.0 REFERENCES

Not applicable.

#### 9.0 APPENDIX

#### 9.1 Criteria for Markedly Abnormal Values

# 9.1.1 Hematology, Serum Chemistry, Vital Signs, and 12-lead ECG (except Upper MAV Criteria of QTcF Interval)

For each parameter, all evaluable data (ie, non-missing data) obtained up to Day 11 will be classified as a MAV or not. The criteria in the table below will be used.

For each parameter and subject, classifications will be made according to the conditions i) to iii) provided below. The lower and the upper criteria will be considered separately.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that doesn't meet the MAV criteria will be considered as a subject without MAV.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV for that parameter.

#### **Hematology**

| | MAV Criteria | |
|---|---|---|
| Parameter | Lower Criteria | Upper Criteria |
| Red blood cells (×10 <sup>12</sup> /L) | <0.8×LLN | >1.2×ULN |
| White blood cells ( $\times 10^9/L$ ) | <0.5×LLN | >1.5×ULN |
| Hemoglobin (g/L) | <0.8×LLN | >1.2×ULN |
| Hematocrit (%) | <0.8×LLN | >1.2×ULN |
| Platelets (×10 <sup>9</sup> /L) | <75 | >600 |
| Neutrophils (%) | <0.5×LLN | >1.5×ULN |
| Eosinophils (%) | - | >2×ULN |
| Basophils (%) | - | >3×ULN |
| Monocytes (%) | - | >2×ULN |
| Lymphocytes (%) | <0.5×LLN | >1.5×ULN |
| aPTT (sec) | | >1.5×ULN |
| PT/INR | | >1.5 |

## **Serum Chemistry**

| | MAV Criteria | |
|----------------------------------|----------------|----------------|
| Parameter | Lower Criteria | Upper Criteria |
| Alanine aminotransferase (U/L) | - | >3×ULN |
| Alkaline phosphatase (U/L) | - | >3×ULN |
| Aspartate aminotransferase (U/L) | - | >3×ULN |
| GGT (U/L) | - | >3×ULN |
| Total bilirubin (μmol/L) | - | >34.2 |
| Direct bilirubin (μmol/L) | - | >2×ULN |
| Creatine kinase (U/L) | - | >5×ULN |
| Albumin (g/L) | <25 | - |
| Total protein (g/L) | <0.8×LLN | >1.2×ULN |
| Uric Acid (mmol/L) | - | >0.773 |
| Triglycerides (mmol/L) | - | >2.5×ULN |
| Glucose (mmol/L) | <2.8 | >19.4 |
| Potassium (mmol/L) | <3.0 | >6.0 |
| Sodium (mmol/L) | <130 | >150 |
| Magnesium (mmol/L) | < 0.5 | >1.2 |
| Calcium (mmol/L) | <1.75 | >2.88 |
| Chloride (mmol/L) | <75 | >126 |
| Amylase (U/L) | - | >2×ULN |
| Serum creatinine (µmol/L) | - | >177 |

## Vital Signs

| | MAV ( | Criteria |
|---------------------------------|----------------|----------------|
| Parameter | Lower Criteria | Upper Criteria |
| Body Temperature (°C) | <35.6 | >37.7 |
| Systolic Blood Pressure (mmHg) | <85 | >180 |
| Diastolic Blood Pressure (mmHg) | <50 | >110 |
| Pulse (bpm) | <50 | >120 |

#### 12-lead ECG

| | MAV ( | MAV Criteria |
|----------------------|----------------|----------------|
| Parameter | Lower Criteria | Upper Criteria |
| Heart Rate (bpm) | <50 | >120 |
| QT Interval (msec) | <=50 | >=460 |
| QTcF Interval (msec) | <=50 | - |

### 9.1.2 12-lead ECG (Upper MAV Criteria of QTcF Interval)

All evaluable data (ie, non-missing data) obtained up to Day 11 will be classified as a MAV or not. The criteria in the table below will be used. Note that the observed value and the change from baseline used for classification should be measurements taken on the same day.

For each subject, classifications will be made according to the conditions i) to iii) provided below.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that meets any of the following will be considered as a subject without MAV.
- Observed value is less than 450 msec and not missing.
- Change from baseline is less than 30 msec and not missing, and observed value is less than 500 msec and not missing.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV.

| | MAV Criteria | |
|---|---|---|
| Parameter | Lower Criteria | Upper Criteria |
| QTcF Interval (msec) | - | If either of the following conditions is met: |
| | • observed value >=500 | |
| | | • change from baseline >= 30 and observed value >=450 |

## TAK-438\_114-Statistical Analysis Plan-2017-08-30

## ELECTRONIC SIGNATURES

| Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH:mm 'UTC') |
|---|---|---|
| PPD | Biostatistics Approval | 04-Sep-2017 01:41 UTC |
| PPD | Clinical Pharmacology Approval | 04-Sep-2017 04:06 UTC |
| PPD | Biostatistics Approval | 04-Sep-2017 13:13 UTC |
| PPD | Clinical Approval | 06-Sep-2017 04:56 UTC |
| PPD | Pharmacovigilance Approval | 19-Sep-2017 12:11 UTC |